CLINICAL TRIAL: NCT02269982
Title: Development of Circulating Molecular Predictors of Chemotherapy and Novel Hormonal Therapy Benefit in Men With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Prospective CiRculating prOstate Cancer Predictors in HighEr Risk mCRPC studY
Acronym: PROPHECY
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Weill Medical College of Cornell University (Other); Johns Hopkins University (Other); Dana-Farber Cancer Institute (Other); Memorial Sloan Kettering Cancer Center (Other); Epic Sciences (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00056936
Record Dates: First submitted 2014-10-09; First posted 2014-10-21 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All 120 subjects will have blood collected at 3 time points for CTC-based AR-v7 analysis. Biopsy samples will be collected from up to 20 consenting subjects who are already undergoing a standard of care metastatic biopsy or from a research only biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- men with mCRPC prior to enzalutamide/abiraterone
  Interventions: Device: AR-v7 assays

INTERVENTIONS:
Device: AR-v7 assays

SUMMARY:
This study will develop a first-in-man CTC-based molecular taxonomy of CRPC in the context of novel AR-directed therapies, categorize different patterns of resistance in this disease setting, and describe their evolution over time and treatment.

DETAILED DESCRIPTION:
The study will construct a multi-center clinical database of men before and after treatment with abiraterone acetate, enzalutamide, and taxane chemotherapy, and will comprehensively analyze CTC DNA for copy gains/losses and whole exome sequencing for acquired mutations, CTC RNA for AR-variants and evidence of epithelial plasticity, and plasma circulating tumor DNA (ctDNA) for whole exome sequencing. Significantly, the investigators will pair the presence of key proposed circulating biomarkers of treatment resistance with patient outcomes on these systemic therapies for the purpose of developing predictive biomarkers that may have direct clinical utility in guiding choice of therapies. It is proposed that specific AR-v's (i.e. AR-v7), biomarkers of epithelial plasticity, and microtubule interacting protein variants will convey docetaxel resistance and be enriched in men failing abiraterone acetate or enzalutamide, while other AR genomic events (AR amplification, AR-v567es, AR mutations, GR overexpression) will be responsive to taxane chemotherapy. This work represents a first-in-field comprehensive analysis of CTC molecular profiles for the development of a CTC molecular taxonomy of mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Pure small cell or neuroendocrine tumors of the prostate are not permitted.
2. Clinical or radiographic evidence of metastatic disease.
3. Planned therapy with either enzalutamide and/or abiraterone acetate within the coming 6 weeks
4. Castrate levels of testosterone (<50 ng/dl) at most recent assessment and/or documented ongoing Androgen Deprivation Therapy for at lease three months.
5. Evidence of disease progression on or following most recent therapy as evidenced by at least one of the following:

   * Radiographic evidence of disease progression as defined by one or more new bone scan lesions that is not consistent with flare/healing, or growth of soft tissue/visceral metastases to greater than one centimeter (cm) in longest diameter (2 cm shortest diameter for lymph nodes).
   * Clinical progression as defined by the treating physician (such as pain progression)
   * Consecutive PSA rises meeting PSA progression criteria as determined by PCWG2 criteria (increase that is >25% and >2 ng/mL above the nadir, and which is confirmed by a second value 3 or more weeks later)
6. At least two of the following high risk features during screening for rapid disease progression:

   1. Anemia with a hemoglobin <12.0 g/dl
   2. Elevated alkaline phosphatase above the institution upper limit of normal
   3. High lactate dehydrogenase (LDH) above the upper limit of normal
   4. Prior therapy with enzalutamide, abiraterone acetate, or orteronel. Patients are not permitted if they are continuing on the same therapy or restarting a therapy that they have been exposed to in the past.
   5. Presence of visceral metastasis on imaging
   6. Presence of clinically significant pain requiring opioid analgesia
   7. Patients with a Cellsearch CTC > 5 cells per 7.5 mL whole blood (if available as standard of care) are eligible without additional high risk features
   8. PSA doubling time under 3 months on most recent therapy
   9. Radiographic progression at entry based on new lesion(s) in bone, soft tissue, or visceral metastases
7. Age > 18 years.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. History of intercurrent or past medical or psychiatric illness that would make participation in a blood drawing protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).
2. Treatment with an anthracycline or mitoxantrone within 1 week of CTC collection
3. Prior docetaxel in the castration resistant metastatic setting. Patients treated with docetaxel for metastatic castration sensitive disease will be eligible.
4. Unwillingness to be followed longitudinally for serial CTC biomarker studies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes men with progressive metastatic castration resistant prostate cancer (mCRPC).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of median progression free survival (PFS) to AR-v7 status | 2 years

SECONDARY OUTCOMES:
Determine the prevalence of defined categories of a molecular taxonomy of mCRPC using CTC biomarkers and correlate each to clinical benefit (PSA response, PFS) | 4 years
Compare levels of circulating epithelial to mesenchymal transition (EMT) and other epithelial plasticity (EP) biomarkers with mCRPC taxonomic categories and clinical outcomes (PSA decline rates, PFS) | 4 years
Determine molecular lesions in CTCs and ctDNA that consistently emerge during enzalutamide and taxane chemotherapy progression in men with mCRPC | 4 years
Correlate specific AR-v7 assays with clinical outcomes (PSA decline rates, PFS) | 4 years
Correlatate other AR-variants with clinical outcomes (PSA decline rates, PFS) | 4 years
Change in neuroendocrine biomarkers during enzalutamide and taxane progression in men with mCRPC | 4 years
Associate high CTC heterogeneity with PFS, OS, and CTC genotype/phenotypes | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Armstrong, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Scher HI, Armstrong AJ, Schonhoft JD, Gill A, Zhao JL, Barnett E, Carbone E, Lu J, Antonarakis ES, Luo J, Tagawa S, Dos Anjos CH, Yang Q, George D, Szmulewitz R, Danila DC, Wenstrup R, Gonen M, Halabi S. Development and validation of circulating tumour cell enumeration (Epic Sciences) as a prognostic biomarker in men with metastatic castration-resistant prostate cancer. Eur J Cancer. 2021 Jun;150:83-94. doi: 10.1016/j.ejca.2021.02.042. Epub 2021 Apr 21. PMID 33894633
- [Derived] Gupta S, Halabi S, Kemeny G, Anand M, Giannakakou P, Nanus DM, George DJ, Gregory SG, Armstrong AJ. Circulating Tumor Cell Genomic Evolution and Hormone Therapy Outcomes in Men with Metastatic Castration-Resistant Prostate Cancer. Mol Cancer Res. 2021 Jun;19(6):1040-1050. doi: 10.1158/1541-7786.MCR-20-0975. Epub 2021 Mar 26. PMID 33771885
- [Derived] Armstrong AJ, Halabi S, Luo J, Nanus DM, Giannakakou P, Szmulewitz RZ, Danila DC, Healy P, Anand M, Rothwell CJ, Rasmussen J, Thornburg B, Berry WR, Wilder RS, Lu C, Chen Y, Silberstein JL, Kemeny G, Galletti G, Somarelli JA, Gupta S, Gregory SG, Scher HI, Dittamore R, Tagawa ST, Antonarakis ES, George DJ. Prospective Multicenter Validation of Androgen Receptor Splice Variant 7 and Hormone Therapy Resistance in High-Risk Castration-Resistant Prostate Cancer: The PROPHECY Study. J Clin Oncol. 2019 May 1;37(13):1120-1129. doi: 10.1200/JCO.18.01731. Epub 2019 Mar 13. PMID 30865549